CLINICAL TRIAL: NCT02317848
Title: PRevalence, Persistence and prOgnostic ValuE of Sleep Apnea Syndrome in Acute Heart Failure.
Acronym: PROVE-SAS-AHF
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: French Cardiology Society (Other)
Collaborators: ResMed Foundation (Other); Henri Mondor University Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: 2014-01
Record Dates: First submitted 2014-11-10; First posted 2014-12-17 (Estimated); Last update posted 2019-08-05 (Actual); Status verified 2019-02

CONDITIONS: Sleep Apnea Syndrome; Heart Failure
Keywords: Diagnosis; prognostic marker; polygraphy; echocardiography; ECG
MeSH Terms: conditions — Sleep Apnea Syndromes; Heart Failure; Disease | interventions — epicatechin gallate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- patients with acute heart failure (Other): polygraphy, echocardiography, ECG during hospitalisation for acute heart failure
  Interventions: Other: polygraphy and ECG

INTERVENTIONS:
Other: polygraphy and ECG — polygraphy and ECG during hospitalisation for acute heart failure to see Persistence of the severity of SAS after 2 months

SUMMARY:
The prevalence of sleep-disordered breathing is common in patients with stable chronic heart failure (up to 83%). Basically, the SAS is divided into two categories: central SAS (CSAS) and obstructive SAS (OSAS). The two can coexist. In patients with CHF, the presence of SAS is associated with higher mortality.

CHF is associated with a high rate of re-hospitalization and significant morbidity and mortality and is considered as a major medical and economic problem. To date, few studies have investigated the prevalence, severity, persistence and the role of SAS during cardiac decompensation. For different pathophysiological considerations, it is assumed that SAS is exacerbated during AHF. Therefore SAS is not conventionally screened during this phase. This assumption has been questioned recently by some studies which showed stability of the type of SAS and its severity between the decompensation episode and the stable HF.

Our hypothesis is that SAS during an AHF episode of CHF will remain stable both in terms of severity and type at three months of decompensation. Thus early polygraphy may be reliable for identifying HF patients with SAS.

DETAILED DESCRIPTION:
Sleep apnea syndrome (SAS) is common in stable chronic heart failure (CHF) (60-83%) and is divided into two main types: central SAS (CSAS) and obstructive SAS (OSAS). Several studies have shown an association between SAS and HF severity and prognosis (Damy T, et al. European journal of heart failure 2012, 14(9):1009-1019).

Acute heart failure (AHF) is one of the major complications of CHF. It is assumed that during AHF, the severity of apnea syndrome increases due to increased capillary pressure and blood volume, reason why it is common to screen for a SAS after but not during the decompensation phase to avoid its overestimation. Unfortunately, this screening is often performed only in specialized centers and requires another stay in hospital.

The assumption that the severity of SAS increases during AHF has been questioned recently by some studies. These studies suggest that the prevalence of SAS and type are similar in the acute decompensated phase or after stabilization of HF regarding SAS severity and type. Interestingly, in the study conducted at Padeletti, including 10 patients who underwent polysomnography control just before or immediately after discharge from the hospital, all measured parameters remained stable overall. Padeletti M, et al. Sleep medicine 2009, 10(3):353-360).

Khayat et al (Khayat RN, et al. Journal of cardiac failure 2009, 15(9):739-746) demonstrates stability of SAS 6 weeks after an episode of decompensation. In this study 395 patients with AHF were included with a mean LVEF of 33%, 75% (298) had a SAS with 57% as obstructive and 18% as central SAS (ref). 100% of patients diagnosed with an obstructive SAS during the decompensation phase remained with it 6 weeks later. For central SAS and on the 12 patients with two polygraphies, 4 were reported to change type of SAS which become obstructive.

This raises the question of the importance of early diagnosis of SAS during hospitalization for AHF to allow a more rapid care management.

The aim of this multicenter study is to assess the prevalence, persistence of SAS at 3 months following decompensation as well as the prognostic value at 1 year. If SAS is stable between the episode of the AHF and the return to a stable CHF, treatment of SAS may potentially be considered during the admission phase. The benefit of the therapeutic management will of course be validated by a clinical trial.

ELIGIBILITY:
Inclusion Criteria:

* Major Patient.
* Acute heart failure (stage II, III Killip) having clinical conditions of the European Society of Cardiology guidelines 2005 (26: 384-416) regardless of LVEF.

Exclusion Criteria:

* Patients who have not given their consent.
* State of cardiogenic shock.
* SAS known and treated.
* Patients who are not affiliated to a French social security.
* Significant myocardial infarction transmural (ST depression) in the last 3 months.
* Important heart surgery in the last 3 months.
* Resynchronization in the last 3 months.
* Any significant changes in drug or therapy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Actual)
Dates: Start 2014-12; Primary Completion 2019-05-29 (Actual); Study Completion 2019-05-29 (Actual)

PRIMARY OUTCOMES:
Persistence of the severity of SAS at the follow visit (AHI> 15). | 2 months after AHF

SECONDARY OUTCOMES:
type of SAS | 2 months after AHF
Echocardiography parameters ECG Holter, biology | 2 months after AHF
Prognostic at 1 year (mortality and rehospitalization for HF) | 2 months after AHF

CONTACTS AND LOCATIONS:
Locations (4):
- France (4):
  - Hôpital Henri Mondor, Créteil
  - Chu Pitie Salpetriere, Paris
  - Hôpital BICHAT, Paris
  - Chu Saint Etienne, Saint-Etienne